CLINICAL TRIAL: NCT03143829
Title: Promoting Cancer Symptom Management in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: University of South Florida (Other); Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R15NR015851-01 (NIH)
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Neoplasms; Chemotherapy-induced Nausea and Vomiting
Keywords: gerontology; symptom self-management; Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Neoplasms; Vomiting

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an intervention or wait control group. The intervention group receives an educational intervention at the start of the study. The wait control group receives the intervention at the end.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): electronic Symptom Self-Management Training- CINV (eSSET-CINV) is an educational intervention administered once at the start of treatment
  Interventions: Other: eSSET-CINV
- Wait Control group (Active Comparator): The Wait control group receives the electronic Symptom Self-Management Training- CINV (eSSET-CINV) at the last study visit. Outcomes will be compared to the Intervention group at the end of the study.
  Interventions: Other: eSSET-CINV

INTERVENTIONS:
Other: eSSET-CINV — This intervention is an educational intervention, a serious game, which allows older adults under treatment for cancer to practice making self-care decisions for an avatar who is being sent home after their first chemotherapy treatment. This serious game is coupled with a discussion with a nurse about choices related to managing nausea and vomiting at home.
  Other Names: Managing at home: CINV

SUMMARY:
The purpose of the project is to estimate the effect size of a technology based intervention for older adults with cancer for nausea and vomiting. Participants will be randomized to either an intervention or a wait control group. Outcomes such as symptom severity, quality of life and resource use will be examined.

DETAILED DESCRIPTION:
The goal of this study is to increase the self-management behaviors for chemotherapy induced nausea and vomiting (CINV) and reduce treatment-related negative outcomes in older adults with cancer. CINV is a common reason for unplanned emergency department and/or hospital admissions in older adults with cancer. Early reinforcement of standard education and reframing preconceived beliefs about the potential serious consequences of CINV and the symptoms ability to be successfully managed will increase effective self-management behaviors and improve patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 65 and older
* newly diagnosed with any cancer
* treatment with any chemotherapeutic agent with a moderate to severe emetic potential (on a 3- or 4- week cycle)
* proficient in English
* have a telephone.

Exclusion Criteria:

* Patients with previous diagnosis and treatment for cancer
* advanced or end stage disease with a palliative intent
* visually or hearing impaired.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Loerzel, PhD, Principal Investigator — University of Central Florida
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from June 2016 through August 2018 at the outpatient treatment center at the cancer center
Period: Overall Study
Arm/Group | Intervention Group | Wait Control Group
Started | 38 | 42
Completed | 33 | 32
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 1 | 1
Not completed — changed treatment, no longer eligible | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait Control Group | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.11 (5.311) | 70.26 (6.012) | 69.71 (5.684)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 42 | 80

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity Change Over Time
Description: Symptom Representation Questionnaire (SRQ)[20] , a 24-item self-report measure will be used to identify presence and severity of common treatment-related symptoms (0-10 Likert scale), including nausea and vomiting (N/V). This measure asks respondents to think about their symptoms over the past week. Higher values indicate a worse outcome
Time Frame: assessed at baseline (week 1), week 4,week 7, week 10. differences between groups at week 10 are being reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait Control Group
Number analyzed (Participants) | 38 | 42
score on a scale | 4.13 (3.240) | 3.81 (3.293)
Statistical Analysis 1: Comparison: Intervention Group vs Wait Control Group; Differences at week 10; Test type: Other; p = 0.083, t-test, 2 sided

2. Primary Outcome: Self-management Behaviors Over Time
Description: An investigator-developed Symptom Management Checklist (SMC) will measure CINV self-management prevention behaviors. Participants will complete this daily at home between chemotherapy cycles. Higher numbers indicate more frequent management.
Time Frame: data was assessed at weeks 4,7, 10, the mean number of behaviors (behaviors) combined at each time point is reported
Measure: Mean (Standard Deviation); unit: Behaviors
Arm/Group | Intervention Group | Wait Control Group
Number analyzed (Participants) | 38 | 42
Behaviors | 3.68 (7.59) | 1.38 (4.48)
Statistical Analysis 1: Comparison: Intervention Group vs Wait Control Group; Descriptive comparison; Test type: Other; p = .099, t-test, 2 sided

3. Primary Outcome: Health-related Quality of Life Change Over Time
Description: The EORTC-30[21] will measure QOL at each treatment cycle. 0-10 scale, higher scores mean better outcome
Time Frame: assessed at baseline (week 1), week 4, week 7, week 10. the difference between groups at week 10 is being reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Wait Control Group
Number analyzed (Participants) | 34 | 32
score on a scale | 5.76 (1.046) | 5.91 (.893)
Statistical Analysis 1: Comparison: Intervention Group vs Wait Control Group; comparison at time 4; Test type: Other; p = .558, t-test, 2 sided

4. Primary Outcome: Resource Use Over Time
Description: Any unplanned Emergency Department or hospital admission will be recorded via participant report. Higher number indicate higher resource use.
Time Frame: assessed at weeks 4,7,10. the total number of admissions was summed across all time points and participants
Measure: Number; unit: admissions
Arm/Group | Intervention Group | Wait Control Group
Number analyzed (Participants) | 38 | 42
admissions | 19 | 11
Statistical Analysis 1: Comparison: Intervention Group vs Wait Control Group; descriptive comparison of resource use; Test type: Other; p = .153, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Group | Wait Control Group
All-Cause Mortality (participants affected / at risk) | 1/38 | 1/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 0/38 | 0/42

LIMITATIONS AND CAVEATS:
Limitations were noted with the Cognitive representation data. Participants in this study had very little nausea and therefore were inconsistent in how and when they completed this instrument making data analysis unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03143829/Prot_SAP_000.pdf